CLINICAL TRIAL: NCT02102451
Title: A Five Year Plan of Enhanced HCV Monitoring, Primary Care-Based Workforce Development, Rapid Scale-up of HCV Treatment and Public Health Policy Action in HIV Positive Individuals Within Australia.
Brief Title: Control and Elimination Within Australia of Hepatitis C From People Living With HIV
Acronym: CEASE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: VHCRP1208
Record Dates: First submitted 2014-03-20; First posted 2014-04-03 (Estimated); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Hepatitis C; HIV; HIV-HCV Coinfection
Keywords: Interferon-free; Direct acting antiviral (DAA); Treatment as prevention; Surveillance; Feasibility
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Dry Blood Spot -whole blood collected on filter paper and dried.
  EDTA Plasma
  Peripheral Blood Mononuclear Cell's (PBMC's)
  Samples will be used for HCV related tests including HCV antibody, HCV RNA and HCV genotypes/sequencing that will be performed at the central laboratory from the research samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate the feasibility of rapid scale-up of new hepatitis C (HCV) treatments, known as interferon-free Direct Acting Antiviral (DAA) drugs, and impact on the proportion of people with HCV within the HIV-HCV coinfected population of Australia.

It is hypothesised that a rapid scale-up of hepatitis C treatment with interferon-free therapies in individuals with HIV-HCV coinfection will assist in controlling HCV infection in this population.

DETAILED DESCRIPTION:
This project has seven major components which will occur independently but are linked to the central theme of controlling and eliminating HCV infection from the majority of the Australian HIV positive population.

Database of HIV-HCV individuals (CEASE-D):

Surveillance of HIV-HCV positive individuals will occur through the enrolment into the CEASE-D observational study database. The proportion with HCV viraemia in this population will be determined through three cross-sectional surveys; at enrolment (2014-2016), follow-up 1 (2017-2018) and follow-up 2 (2019-2020). Participation will involve providing informed consent, collection of limited clinic and demographic information, a dried blood spot sample, patient completed CEASE questionnaires and FibroScan® (where available). It is estimated that approximately 1000 HIV-HCV coinfected individuals will be enrolled into the CEASE-D database.

Modelling (CEASE-M):

Mathematical modeling will be undertaken to examine various treatment strategies, including HCV treatment scale-up timelines. The data from the first cross-sectional survey of the HCV surveillance phase (CEASE-D) will inform components of the modeling.

HCV Education for HIV prescribers (CEASE-E):

A comprehensive education program in HCV treatment with interferon-free DAA therapy will be conducted with HIV prescribers with high HCV caseloads in preparation for the rapid scale-up of HCV treatment.

HCV Treatment Scale-Up (CEASE-T):

HCV treatment scale-up with PBS listed regimens will involve primary and tertiary clinics. All patients who are commencing HCV treatment will be invited to participate in CEASE-T which will involve data collection regarding treatment with PBS listed regimens. The regimen and duration will be determined by the treating clinician according to PBS prescribing guidelines. At selected sites subjects will be offered enrollment into a more intensive follow-up substudy (I-STEP) involving collection of research EDTA plasma samples, patient completed behavioural questionnaires and FibroScan® (where available). Patients with recurrent viraemia during or following treatment (relapse/reinfection) may also be entered into a separate substudy cohort (CEASE-V)

Recurrent Viraemia Treatment (CEASE-V) At selected sites patients with on-treatment virological failure (nonresponse or viral breakthrough) or post-treatment recurrent viraemia (relapse or reinfection) will be entered into an intensive follow-up cohort (CEASE-V). Participation will involve providing informed consent, collection of research EDTA plasma samples and patient completed behavioural questionnaires. Patients may be offered retreatment with PBS listed regimens. The decision to retreat as well as the regimen and duration will be determined by the treating clinician according to PBS prescribing guidelines.

Dried Blood Spot Validation Sub-study (DBS Sub-study) At selected sites patients will be invited to participate in the Dried Blood Spot Validation Sub-study (DBS Sub-study). HIV/HCV study participants and HCV control participants will be mailed DBS self-collection kits and questionnaires to evaluate feasibility, acceptability and validity of self-collected DBS samples compared to clinic collected plasma samples. Pre and post DBS acceptability questionnaires will be completed.

Qualitative Sub-study (CEASE-Q) At selected sites patients will be invited to participate in the Qualitaitive Sub-study (CEASE-Q). Semi-structured interviews will be used to explore risk behaviour pre and post DAA therapy, participant experience of DAA therapy and, in untreated participants, facilitators and barriers to DAA therapy.

ELIGIBILITY:
Inclusion Criteria:

CEASE-D:

1. 18 years of age or older
2. Voluntarily signed the informed consent form
3. HIV positive
4. HCV antibody positive
5. Adequate English and mental health status to provide written informed consent and comply with study procedures

CEASE-T (ISTEP):

1. 18 years of age or older
2. Voluntarily signed the informed consent form
3. HIV positive
4. HCV RNA positive
5. Adequate English and mental health status to provide written informed consent and comply with study procedures
6. Undergoing DAA therapy HCV treatment.

CEASE-V:

1. 18 years of age or older
2. Voluntarily signed the informed consent form
3. HIV positive
4. Undergone IFN-free DAA therapy for HCV

6) On treatment virological failure or post-treatment recurrent viraemia as defined by either:

1. Non-response: Failure of viral suppression on IFN-free DAA therapy
2. Virological breakthrough on IFN-free DAA therapy
3. Post-treatment recurrent viraemia: Detectable HCV RNA post-treatment following an end-of-treatment response (ETR, undetectable HCV RNA at end of treatment)

   DBS Sub-study Population:

   1) 18 years of age or older 2) Voluntarily signed the informed consent form 3) HIV positive 4) HCV antibody positive 5) Adequate English and mental health status to provide written informed consent and comply with study procedures 6) Under follow-up within I-STEP post-treatment for HCV

   DBS Sub-study Controls:

   1) 18 years of age or older 2) Voluntarily signed the informed consent form 3) HIV negative 4) HCV antibody positive 5) Undergoing DAA therapy for HCV and requiring confirmation of SVR post therapy 6) Adequate English and mental health status to provide written informed consent and comply with study procedures

   CEASE-Q:

   1) 18 years of age or older 2) Voluntarily signed the informed consent form 3) HIV positive 4) HCV antibody positive 5) Adequate English and mental health status to provide written informed consent and comply with study procedures 6) Under follow-up within I-STEP post-treatment for HCV

   Exclusion Criteria:

   CEASE-D:

   1) Inability or willingness to comply with protocol requirements

   CEASE-T:

   1) Inability or willingness to comply with protocol requirements

   CEASE-V:

   1) Inability or willingness to comply with protocol requirements

   DBS Sub-study:

   1) Inability or willingness to comply with protocol requirements

   CEASE-Q:

   1) Inability or willingness to comply with protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults living with HIV-HCV coinfection
Sampling Method: Probability Sample
Enrollment: 492 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
HCV viraemia | 5 years
  Proportion of HCV viraemia within the Australian HIV-HCV population over a five year period

SECONDARY OUTCOMES:
Needs, behaviour and attitudes towards HCV treatment | 5 years
  To assess the needs, risk behaviour and willingness to undergo treatment in HIV-HCV coinfected individuals
HCV treatment uptake | 5 years
  To monitor levels and types of HCV treatment uptake over time as therapies for HCV infection evolve
Factors associated with HCV treatment and retreatment | 5 years
  To examine factors which are associated with treatment and retreatment uptake at the tertiary, secondary and primary care level, including the influence of liver stage disease, genotype and availability of treatment regimens on treatment decision making
HCV treatment response rates | 5 years
  To assess treatment response rates to the roll out of interferon-free DDA therapies including the reasons for treatment failure
Rates of HCV retreatment | 5 years
  To monitor rates of retreatment including for treatment failure and for reinfection
HCV transmission history | 5 years
  To characterise, using molecular epidemiology, HCV transmission history within the HIV-HCV coinfected population

CONTACTS AND LOCATIONS:
Overall Officials: Gail Matthews, MbChB, MRCP, FRACP, PhD, Principal Investigator — Kirby Institute, University of New South Wales; Greg Dore, BSc, MBBS, FRACP, MPH, PhD, Principal Investigator — Kirby Institute, University of New South Wales
Locations (18):
- Australia (18):
  - Dr Doong's Surgery, Burwood, New South Wales
  - Blue Mountains Sexual Health and HIV Centre, Katoomba, New South Wales
  - Sydney Sexual Health Centre, Sydney, New South Wales
  - East Sydney Doctors, Sydney, New South Wales
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - Kirketon Road Centre, Sydney, New South Wales
  - St Vincent's Hospital, Sydney, New South Wales
  - Taylor Square Private Clinic, Sydney, New South Wales
  - The Albion Centre, Sydney, New South Wales
  - Western Sydney Sexual Health, Sydney, New South Wales
  - Nepean Sexual Health and HIV Clinic, Sydney, New South Wales
  - Brisbane Sexual Health Clinic, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Melbourne Sexual Health Centre, Carlton, Victoria
  - Northside Clinic, Fitzroy North, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Prahran Market Clinic, Prahran, Victoria
  - The Centre Clinic, St Kilda, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinello M, Carson JM, Post JJ, Finlayson R, Baker D, Read P, Shaw D, Bloch M, Doyle J, Hellard M, Filep E, Hosseini-Hooshyar S, Dore GJ, Matthews GV. Control and Elimination of Hepatitis C Virus Among People With HIV in Australia: Extended Follow-up of the CEASE Cohort (2014-2023). Open Forum Infect Dis. 2024 Dec 17;11(12):ofae665. doi: 10.1093/ofid/ofae665. eCollection 2024 Dec. PMID 39691290
- [Derived] Martinello M, Yee J, Bartlett SR, Read P, Baker D, Post JJ, Finlayson R, Bloch M, Doyle J, Shaw D, Hellard M, Petoumenos K, Lin L, Marks P, Applegate T, Dore GJ, Matthews GV. Moving Towards Hepatitis C Microelimination Among People Living With Human Immunodeficiency Virus in Australia: The CEASE Study. Clin Infect Dis. 2020 Sep 12;71(6):1502-1510. doi: 10.1093/cid/ciz985. PMID 31585005